CLINICAL TRIAL: NCT00000749
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of 200 Mcg of gp120 (CHO) BIOCINE in MF59 Emulsion Versus the Emulsion Control: Three Injections at 0, 1, and 6 Months
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Biocine (Industry)
Model: Parallel | Purpose: Prevention
Other Study IDs: AVEG 007C
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: rgp120/HIV-1 SF-2

SUMMARY:
To evaluate in healthy volunteers the safety and immune response to 200 mcg gp120 candidate vaccine in MF59 emulsion without MTP-PE at 0, 1 and 6 months.

Preliminary evaluations of two dose levels of gp120 administered to volunteers in protocol VEU 007A indicate that a gp120 dose of potentially greater immunogenicity may be of interest.

DETAILED DESCRIPTION:
Preliminary evaluations of two dose levels of gp120 administered to volunteers in protocol VEU 007A indicate that a gp120 dose of potentially greater immunogenicity may be of interest.

Ten healthy volunteers receive 200 mcg gp120 in MF59 emulsion, and four volunteers receive placebo consisting of MF59 emulsion in PBS vehicle. Injections are given at months 0, 1, and 6. Patients are followed for 12 months following the third injection.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* Negative ELISA for HIV.
* Normal cell-mediated immune responses using Merieux skin test.
* Normal urinalysis.

Exclusion Criteria

Co-existing Condition:

Subjects with the following conditions are excluded:

* Evidence of psychological or psychiatric problems that may lead to noncompliance with study requirements.
* Positive syphilis serology. If serology is documented as a false positive or is due to a remote (> 6 months) treated infection, subject is eligible.
* Circulating hepatitis B surface antigen.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications.
* History of anaphylaxis or other adverse reactions to vaccines.

Prior Medication:

Excluded:

* Prior HIV vaccines.
* Immunoglobulins or vaccines within the past 3 months.
* Experimental agents within the past 30 days.

Prior Treatment:

Excluded:

* Blood transfusions or cryoprecipitates within the past 3 months.

Identifiable high-risk behavior for HIV infection, including:

* Any history of intravenous (IV) drug use within the past year.
* Syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease) in the past 6 months.
* More than two sexual partners, or sexual contact with a high-risk partner, in the past 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14

CONTACTS AND LOCATIONS:
Overall Officials: Graham B, Study Chair
Locations (2):
- United States (2):
  - Vanderbilt Univ Hosp, Nashville, Tennessee
  - Univ of Washington / Pacific Med Ctr, Seattle, Washington